CLINICAL TRIAL: NCT06919835
Title: CiLostAzol for pReventIon of Recurrent sTroke in Africa
Acronym: CLARITY-Africa
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Responsible Party: Principal Investigator, Bruce Ovbiagele, Chief of Staff, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-41599
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke; Africa; post-stroke
MeSH Terms: conditions — Stroke | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cilostazol Experimental Arm (Experimental): Patients allocated to the experimental arm will receive 100mg of cilostazol tablets taken twice daily. To mitigate side-effects in both treatment arms, all patients will begin one tablet daily and titrate to the full dose (one tablet twice daily) after 2 weeks. Participants will stay on the full dose of cilostazol for the remainder of the study.
  Interventions: Drug: Cilostazol 100 mg
- Control Arm (No Intervention): Standard of post-stroke care

INTERVENTIONS:
Drug: Cilostazol 100 mg — Patients allocated to the experimental arm will receive 100mg of cilostazol tablets taken twice daily. To mitigate side-effects in both treatment arms, all patients will begin one tablet daily and titrate to the full dose (one tablet twice daily) after 2 weeks. Participants will stay on the full dose of cilostazol for the remainder of the study.
  Arms: Cilostazol Experimental Arm

SUMMARY:
Global estimates suggest that sub-Saharan Africa (SSA) now has the highest incidence, prevalence, and worst survival outcomes of stroke. With an estimated 1.4 million stroke survivors, outcomes of stroke in SSA are abysmal with 1-month case fatality at 30% and 3-year mortality rate of 84%. Stroke survivors in Africa are at an inordinately high (and worsening) risk of adverse outcomes including recurrent stroke and cardiac events over the medium- to longterm. Given the paucity of resources in the region, testing of therapies, which are potentially highly clinically efficacious and cost-effective, while developing local stroke research capacity and contributing to the global secondary stroke prevention evidence base, is urgently needed. Cilostazol, a phosphodiesterase 3 inhibitor, has shown promising efficacy and safety mainly among an Asian population by cutting risk of major adverse cardiovascular events including stroke, in half, when added to aspirin or clopidogrel (8% vs. 4%, HR 0.52, 95% CI 0.35-0.77), with no increased risk in bleeding or serious adverse events. Cilostazol's potentially strong efficacy, presumed pleiotropic effects, and relatively low cost, make it a highly appealing agent for use in stroke-prone, low-resource settings. Therefore, the overall objective of the CiLostAzol for pReventIon of recurrent sTroke in Africa (CLARITY-AFRICA) study is to deploy a hybrid study design to demonstrate the efficacy and safety of cilostazol twice daily in reducing MACE over 24 months vs. placebo among 1100 recent stroke patients encountered at 12 hospitals in Ghana. Secondly, CLARITY-AFRICA also seeks to develop an implementation strategy for routine integration and policy adoption of cilostazol for post-stroke cardiovascular risk reduction in an under-resourced system. Given its compelling efficacy among a predominantly Asian population, the National Institute of Neurological Disorders and Stroke (NINDS) is poised to fund a US-based clinical trial to assess the longer-term efficacy and safety of cilostazol in a study titled CiLostAzol for pReventIon of recurrent sTroke (CLARITY). The investigators are also aware that European and Australian funding agencies are considering stroke trials of cilostazol. A concurrently executed CLARITYAfrica trial would allow recruitment of a historically underrepresented and high-risk group (Africans), test a therapy that if efficacious could be affordable for broader regional implementation, permit transcontinental mentorship/collaborations, and leverage NINDS impending investment. CLARITY-AFRICA will assess implementation outcomes such as adoption, acceptability, cost, pertinent to uptake of cilostazol in Ghana to inform policy. Regardless of its outcome, findings from CLARITYAFRICA will contribute meaningful information from the African perspective to inform the formulation of guidelines for global adoption of cilostazol into routine care for secondary CVD risk prevention by international bodies such as the World Health Organization. This application will focus on the first 2 aims of CLARITY-AFRICA to conduct the trial and assess secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Above the age of 30 years; male or female (sex is a biological variable of interest)
2. Ischemic stroke or high-risk TIA (ABCD2 score >= 6) diagnosis no greater than six months before enrollment. Ischemic strokes including lacunar, large vessel atherosclerotic, embolic stroke of undetermined source subtypes are eligible (Ischemic stroke or TIA should be confirmed by either with a cranial CT or MRI within 10 days of symptom onset)
3. Aspirin or clopidogrel monotherapy
4. Subjects with stroke may present with two or more of the following additional conditions: age ≥65 years, documented diabetes mellitus or previous treatment with oral hypoglycemic or insulin; documented hypertension >140/90mmHg or previous treatment with anti-hypertensive medications; Mild to moderate renal dysfunction (eGFR 60-30ml/min/1.73m2); Prior myocardial infarction
5. Legally competent to sign informed consent or have a LARs who is able to provide consent for them
6. In the opinion of the treating physician, patient is medically stable, capable of participating in a randomized trial, and willing and able to attend follow-up.
7. Able to do labs at all study intervals (7 visits total)

Exclusion Criteria:

1. Unable to provide a valid informed consent
2. Contraindications to cilostazol (namely (i) hypersensitivity, (ii) active pathologic bleeding, e.g. bleeding peptic ulcer, intracranial bleeding due to reversible platelet aggregation, (iii) congestive cardiac failure.)
3. Hemorrhagic stroke survivor within the last 2 years
4. Use of an anticoagulant medication or indication for use of an anticoagulant (e.g. atrial fibrillation)
5. On dual antiplatelet therapy (patients are eligible after completion of a course of dual antiplatelet therapy)
6. Modified Rankin Scale 5
7. Thrombocytopenia (platelet count <1000,000)
8. Severe liver dysfunction (active hepatitis or hepatic insufficiency with Child-Pugh score B or C)
9. Congestive heart failure, defined as NYHA Class III or above (marked limitation of physical activity)
10. Nursing/pregnant mothers

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants with Major Adverse Cardiovascular Events | 36 months

SECONDARY OUTCOMES:
Percent of Participants with of Major and Minor bleeding | 24 months
Percent of Participants with Recurrent stroke (Ischemic or Hemorrhagic) | 24 months
Percent of Participants with Cardiovascular Deaths | 24 months
Percent of Participants with All Cause Mortality | 24 months
Neuro-QoL (Quality of Life) | 24 months
  12 monthly
  Neuro-QoL uses T-scores, which are standardized scores:
  Mean (average) = 50 Standard deviation = 10
  Interpreting T-scores:
  Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
  For negative domains (e.g. anxiety, depression, fatigue):
  Higher = Worse
  We will compare mean Neuro-QoL scores between the two arms of the study at study completion as well as proportions with mild, moderate and severe impairment.
Exploratory outcomes Montreal Cognitive Assessment | 24 months
  6 monthly. Comparison of Slopes of MOCA scores over 24 months. Range of scores on MOCA: 0 to 30.
  MOCA screening tool is used to detect mild cognitive impairment and early signs of dementia. It evaluates several cognitive domains, including:
  Memory Attention Language Visuospatial skills Executive function Orientation
  A score of 26 or above is considered normal. Scores below 26 may suggest cognitive impairment, depending on education level and clinical context.
Quality of Life (EQ-5D Questionnaire) | 24 months
  The EQ-5D is a health-related quality of life questionnaire with two parts:
  Descriptive system: Assesses 5 dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each rated on 3 or 5 levels (from no problems to extreme problems).
  Visual Analog Scale (VAS): Rates overall health from 0 (worst) to 100 (best).
  Scoring:
  The 5-digit health state is converted into a summary index score (range: <0 to 1), with 1 = full health.
  The VAS reflects the person's self-rated health.
  We will compare scores between the two arms at study completion.
Modified Rankin Score | 24 months
  The Modified Rankin Scale (mRS) measures the degree of disability or dependence in daily activities after a stroke or other neurological injury.
  Scoring:
  0 - No symptoms
  1. - No significant disability; able to carry out all usual activities
  2. - Slight disability; unable to do all previous activities but able to look after own affairs
  3. - Moderate disability; needs some help but can walk unassisted
  4. - Moderately severe disability; unable to walk or attend to bodily needs without help
  5. - Severe disability; bedridden, incontinent, requires constant care
  6. - Dead

CONTACTS AND LOCATIONS:
Locations (1):
- Kwame Nkrumah University of Science & Technology, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No
Individual participant level data will be aggregated and maintained as de-identified to protect PHI